CLINICAL TRIAL: NCT03667924
Title: Utilizing Senior Companions to Enhance Dementia Care Services and Supports
Brief Title: Utilizing Senior Companions to Enhance Dementia Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Johns Hopkins University (Other); Brown University (Other); National Institute on Aging (NIA) (NIH); University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004176; R61AG061903 (NIH)
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Caregiving; Community-based care; Long-term services and supports; Volunteer
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Enrollment: Number of participants: 44 (33 senior volunteers; 7 clients (PWML); 4 caregivers)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PorchLight Project Intervention Group (Experimental): Participants in the intervention group will receive home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
  Interventions: Behavioral: PorchLight Project

INTERVENTIONS:
Behavioral: PorchLight Project — Senior Companions (or other LSS-MN volunteers providing senior companionship services) who deliver the PorchLight Project will complete online CARES® Dementia Care Specialist training modules, additional trainings delivered by the research team (1. overview of the PorchLight Project, 2. review of the National Consensus Guidelines on Palliative Care, 3. review of the list of guided questions, and 4. review of journaling approach and LTSS resources), and participate in unstructured monthly check-ins (discussions and case review as applicable) with the research team.

SUMMARY:
The inability of healthcare systems to effectively manage Alzheimer's disease and related dementias (ADRD) often results in families remaining unaware of important community-based, long-term services and supports (LTSS) that could help to mitigate the negative effects of cognitive impairment. This project will feature a collaboration between Lutheran Social Service of Minnesota and the University of Minnesota to evaluate a novel adaption of the volunteer Senior Companion Program (SCP) to: a) assist families better manage ADRD at home; b) identify and facilitate the use of LTSS; and c) improve engagement with primary care providers throughout the state of Minnesota. If successful, the PorchLight Project will offer a potentially efficient, wide-ranging service model for states and communities to implement for persons with ADRD and their caregiving families.

DETAILED DESCRIPTION:
This project will evaluate a novel adaption of the Senior Companion Program (SCP) administered by Lutheran Social Service of Minnesota to assist families better manage their relatives' Alzheimer's disease or related dementias (ADRDs); identify and facilitate use of community-based long-term services and supports (LTSS); and improve engagement with healthcare providers. This intervention, called the PorchLight Project has the following aims:

Specific Aim 1. Implement PorchLight Project for 25 persons with ADRD or memory concerns (collectively, persons with memory loss [PWML]) and/or their caregivers in one urban and rural region of Minnesota. A convergent parallel mixed methods design [(QUAN+QUAL)-->QUAL] will be utilized to examine the feasibility, acceptability, and utility of PorchLight Project for 25 families and their SC-Ds (n = 20) over a 3-month period (i.e., Stage I of the NIH Stage Model).

Specific Aim 2. Refine PorchLight Project delivery and implementation for efficacy evaluation. Activities to support this aim will include assessment of R61 milestones and incorporation of R61 findings to refine the PorchLight Project prior to efficacy evaluation. Through stakeholder engagement with the Dementia Healthcare Research Advisory Group (DHR) as well as analysis of the various quantitative and qualitative data elements collected during this Phase, we will finalize and refine effective training approaches for PorchLight Project Senior Companions (SCs), identify and confirm stakeholder-centric measures, and enhance the overall implementation of the PorchLight Project to inform a subsequent R33 Phase.

ELIGIBILITY:
Inclusion criterion for the Senior Companion: 1) be a current volunteer through LSS-MN 2) be willing to complete the CARES® modules and 4-part training session provided by UMN research staff and 3) be 21 years of age or older.

Inclusion criteria for the PWML will be based on one of the following scenarios: 1) the person or their caregiver are concerned about the person's memory loss, 2) the person has a physician diagnosis of ADRD, 3) the caregiver (or PWML) scores 2 or greater on the AD8. The PWML must be 55 years of age or older.

Inclusion criteria for the caregiver is that the individual is 1) 21 years of age or older, 2) self-identifies as someone who provides help to the PWML because of their cognitive impairments, and 3) the care recipient is eligible for the study as per the above criteria.

Exclusion Criteria:

A PWML or caregiver will be ineligible if they have a diagnosis of a serious psychiatric illness, their symptoms have worsened in the last 6 months, and they don't receive steady, ongoing treatment for those symptoms.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosebush CE, Stabler H, Nkimbeng M, Louwagie K, Fields NL, Jutkowitz E, Shippee TP, Gaugler JE. The Porchlight Project: A Pilot Study to Adapt the Senior Companion Program to Enhance Memory Care Services and Supports. Gerontol Geriatr Med. 2021 May 14;7:23337214211017651. doi: 10.1177/23337214211017651. eCollection 2021 Jan-Dec. PMID 34036120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From PMCID: PMC8127785/PMID: 34036120: "Regional program coordinators (RPCs) introduced the PorchLight Project to volunteers during SCP meetings and via telephone...Enrolled volunteers assisted RPCs in recruiting clients and caregivers by distributing flyers and permission to contact forms during their usual visits; RPCs and lead volunteers followed up via telephone as needed."
Pre-assignment Details: Not applicable; as this was a single arm pilot study, all enrolled participants were assigned to the Porchlight Project group.
Groups:
- PorchLight Project Intervention Group: Clients: Clients in the intervention group received home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
- Porchlight Project Intervention Group: Volunteers: PorchLight Project: Senior Companions (or other LSS-MN volunteers providing senior companionship services) who delivered the PorchLight Project completed online CARES® Dementia Care Specialist training modules, additional trainings delivered by the research team (1. overview of the PorchLight Project, 2. review of the National Consensus Guidelines on Palliative Care, 3. review of the list of guided questions, and 4. review of journaling approach and LTSS resources), and participated in unstructured monthly check-ins (discussions and case review as applicable) with the research team.
- Porchlight Project Intervention Group: Caregivers: If caregivers were available and/or lived with clients, caregivers also received home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
Period: Baseline Completed
Arm/Group | PorchLight Project Intervention Group: Clients | Porchlight Project Intervention Group: Volunteers | Porchlight Project Intervention Group: Caregivers
Started | 7 | 33 | 4
Completed | 7 | 31 | 4
Not Completed | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Period: 1-month Completed/Training (Volunteers)
Arm/Group | PorchLight Project Intervention Group: Clients | Porchlight Project Intervention Group: Volunteers | Porchlight Project Intervention Group: Caregivers
Started | 7 | 31 | 4
Completed (Please note: volunteers did not complete 1-month surveys as did clients and caregivers; instead, the numbers entered here reflect the milestone "training completed") | 6 | 15 | 3
Not Completed | 1 | 16 | 1
Not completed — One client was hospitalized; | 1 | 0 | 0
Not completed — Did not complete full training | 0 | 16 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: 3-month/Volunteers Who Enrolled Clients
Arm/Group | PorchLight Project Intervention Group: Clients | Porchlight Project Intervention Group: Volunteers | Porchlight Project Intervention Group: Caregivers
Started | 6 | 15 | 3
Completed | 5 | 5 | 3
Not Completed | 1 | 10 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Few clients had memory loss, thus only 5 of 15 volunteers were able to apply their training | 0 | 10 | 0
Period: Post-study Interview Completed
Arm/Group | PorchLight Project Intervention Group: Clients | Porchlight Project Intervention Group: Volunteers | Porchlight Project Intervention Group: Caregivers
Started | 5 | 5 | 3
Completed | 5 | 4 | 3
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Note that 33 volunteers were enrolled, and 31 volunteers completed a baseline survey.
Groups:
- PorchLight Project Intervention Group: Clients; Porchlight Project Intervention Group: Volunteers; Porchlight Project Intervention Group: Caregivers: Participants in the intervention group will receive home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
  PorchLight Project: Senior Companions (or other LSS-MN volunteers providing senior companionship services) who deliver the PorchLight Project will complete online CARES® Dementia Care Specialist training modules, additional trainings delivered by the research team (1. overview of the PorchLight Project, 2. review of the National Consensus Guidelines on Palliative Care, 3. review of the list of guided questions, and 4. review of journaling approach and LTSS resources), and participate in unstructured monthly check-ins (discussions and case review as applicable) with the research team.
- Total: Total of all reporting groups
Arm/Group | PorchLight Project Intervention Group: Clients | Porchlight Project Intervention Group: Volunteers | Porchlight Project Intervention Group: Caregivers | Total
Number analyzed (Participants) | 7 | 31 | 4 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.4 (4.7) | 69.7 (7.4) | 60.0 (5.1) | 71.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 25 | 4 | 34
  Male | 2 | 6 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 30 | 4 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 31 | 4 | 35
  White | 7 | 0 | 0 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 31 | 4 | 42
Education: Bachelor's degree or higher [Count of Participants; unit: Participants] | 0 | 10 | 1 | 11
Marital status: Currently married [Count of Participants; unit: Participants] | 2 | 14 | 3 | 19
Employment status: Currently working full- or part-time [Count of Participants; unit: Participants] | 0 | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Utilization of LTSS by PWML and Caregivers
Description: Community-based service utilization of PWML and caregivers will be assessed by asking participants to identify (from a fixed list of options) fifteen different home and community-based services (HCBS).
Time Frame: Baseline, 1-month, 3-month
Population: Analysis population is the same as those who were enrolled, completed a baseline survey, and remained in the study for the 3 month follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Porchlight Project Intervention Group: Clients: Clients in the intervention group will receive home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
- Porchlight Project Intervention Group: Caregivers: If available/present, caregivers in the intervention group will receive home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
Arm/Group | Porchlight Project Intervention Group: Clients | Porchlight Project Intervention Group: Caregivers
Number analyzed (Participants) | 7 | 4
Participants
  Baseline : Case Management | 1 | 1
  Baseline : Visiting nurse services | 2 | 1
  Baseline : Physical therapy | 3 | 2
  Baseline : Speech/Occupational therapy | 1 | 1
  Baseline : Transportation to health services | 2 | 0
  Baseline : Adaptive/assistive supplies | 6 | 2
  Baseline : Social/adult day services | 0 | 0
  Baseline : Congregate meals | 1 | 1
  Baseline : Companion services | 6 | 4
  Baseline : Support group | 0 | 0
  Baseline : In-home respite | 0 | 1
  Baseline : Home delivered meals | 1 | 1
  Baseline : Homemaker/housekeeping | 6 | 3
  Baseline : Live-in paid caregiver | 3 | 1
  Baseline : Education/training services | 0 | 0
  1-month : Case Management: number analyzed (Participants) | 6 | 4
  1-month : Case Management | 2 | 2
  1-month : Visiting nurse services | 3 | 2
  1-month : Physical therapy | 2 | 1
  1-month : Speech/Occupational therapy | 1 | 1
  1-month : Transportation to health services | 2 | 0
  1-month : Adaptive/assistive supplies | 4 | 2
  1-month : Social/adult day services | 0 | 2
  1-month : Congregate meals | 1 | 0
  1-month : Companion services | 6 | 2
  1-month : Support group | 0 | 0
  1-month : In-home respite | 0 | 0
  1-month : Home delivered meals | 0 | 1
  1-month : Homemaker/housekeeping | 4 | 2
  1-month : Live-in paid caregiver | 3 | 1
  1-month : Education/training services | 0 | 0
  3-month : Case Management | 1 | 3
  3-month : Visiting nurse services | 2 | 1
  3-month : Physical therapy | 2 | 1
  3-month : Speech/Occupational therapy | 1 | 1
  3-month : Transportation to health services | 0 | 1
  3-month : Adaptive/assistive supplies | 2 | 1
  3-month : Social/adult day services | 0 | 1
  3-month : Congregate meals | 1 | 1
  3-month : Companion services | 4 | 2
  3-month : Support group | 0 | 0
  3-month : In-home respite | 1 | 0
  3-month : Home delivered meals | 1 | 1
  3-month : Homemaker/housekeeping | 3 | 1
  3-month : Live-in paid caregiver | 1 | 0
  3-month : Education/training services | 0 | 0

2. Primary Outcome: Quality of Primary Care Interactions
Description: A 3-item measure of quality of interaction during primary care provider encounters. The total mean of item-responses was calculated, with a minimum value of 1 and a maximum value of 4. The higher scores mean higher quality interactions.
Time Frame: Baseline, 1-month, 3-month
Population: One participant was loss to follow-up; in addition, at 3 months, one participant indicated they did not attend a doctor's appointment with the care recipient and thus did not complete the subsequent 3-item measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Porchlight Project Intervention Group: Caregivers: If available, caregivers in the intervention group will receive home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
Arm/Group | Porchlight Project Intervention Group: Caregivers
Number analyzed (Participants) | 4
score on a scale
  Baseline | 2.92 (0.83)
  1-Month: number analyzed (Participants) | 3
  1-Month | 3.22 (0.51)
  3-month: number analyzed (Participants) | 2
  3-month | 3.50 (0.71)

3. Primary Outcome: Caregiver Distress: Burden
Description: Caregiver distress will be ascertained with the 22-item Zarit Burden Interview. Scores were summed; the higher the score, the more burden perceived. Minimum score of 0, high score of 88.
Time Frame: Baseline, 1-month, 3-month
Population: One caregiver was lost to follow-up at the 1- and 3-month intervals.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Porchlight Project Intervention Group: Caregivers
Number analyzed (Participants) | 4
score on a scale
  Baseline | 20.5 (18.91)
  1-month: number analyzed (Participants) | 3
  1-month | 30.33 (20.03)
  3-months: number analyzed (Participants) | 3
  3-months | 13.00 (7.00)

4. Primary Outcome: Caregiver Distress: Depressive Symptoms
Description: Caregiver distress will be ascertained with the 20-item Center for Epidemiological Studies-Depression scale. An average/mean, total score of item-responses was computed, with a minimum score of 1 and a high score of 4. The higher the score, the more depressive symptoms experienced.
Time Frame: Baseline, 1-month, 3-month
Population: One caregiver was lost to follow up during the 3 month study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Porchlight Project Intervention Group: Caregivers
Number analyzed (Participants) | 4
score on a scale
  Baseline | 1.29 (0.25)
  1 Month: number analyzed (Participants) | 3
  1 Month | 1.22 (0.19)
  3 Month: number analyzed (Participants) | 3
  3 Month | 1.17 (0.16)

5. Primary Outcome: PWML Well-being
Description: We will assess the PWML health related quality of life using the EQ-5D-5L Visual Analog Scale. The measure is single score of a minimum of 0 and maximum of 100. Higher scores indicate better health.
Time Frame: Baseline, 1-month, 3-month
Population: Two clients were lost to follow-up/did not have longitudinal data available over the 3-month study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Porchlight Project Intervention Group: Clients
Number analyzed (Participants) | 7
score on a scale
  Baseline | 60.71 (23.71)
  1 Month: number analyzed (Participants) | 6
  1 Month | 53.83 (24.46)
  3 Month: number analyzed (Participants) | 5
  3 Month | 52.00 (13.51)

6. Primary Outcome: PWML Depression
Description: PWML Depression will be ascertained using the 15-item Geriatric Depression Scale Short Form. The scale score is summed, with a minimum score of 0 and a maximum of 15. The higher the score, the greater the depressive symptoms experienced/indicated.
Time Frame: Baseline, 1-month, 3-month
Population: Two clients were lost to follow-up during the 3-month study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Porchlight Project Intervention Group: Clients
Number analyzed (Participants) | 7
score on a scale
  Baseline | 4.00 (3.87)
  1-month: number analyzed (Participants) | 6
  1-month | 3.83 (2.86)
  3-month: number analyzed (Participants) | 5
  3-month | 5.00 (3.94)

7. Primary Outcome: PWML Quality of Life
Description: PWML Quality of Life will be ascertained using the 13-item Quality of Life Alzheimer's Disease-Measure (QOL-AD). The measure score is summed. The minimum score is 13 and the maximum score is 52. The higher the score, the greater perceived quality of life.
Time Frame: Baseline, 1-month, 3-month
Population: Two clients were lost to follow-up during the study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Porchlight Project Intervention Group: Clients
Number analyzed (Participants) | 7
score on a scale
  Baseline | 34.86 (8.75)
  1-Month: number analyzed (Participants) | 6
  1-Month | 34.67 (8.31)
  3-Month: number analyzed (Participants) | 5
  3-Month | 37.20 (2.39)

8. Secondary Outcome: Caregiver Self-efficacy
Description: An 8-item measure of caregiver self-efficacy developed by Fortinsky et al. (2002). The score is summed; the higher the score, the more self-efficacy the caregiver perceives. The minimum score on the scale is 8, the maximum is 40.
Time Frame: Baseline, 1-month, 3-month
Population: One caregiver was lost to follow-up over the 3-month study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Porchlight Project Intervention Group: Caregivers
Number analyzed (Participants) | 4
score on a scale
  Baseline | 32.00 (2.71)
  1-month: number analyzed (Participants) | 3
  1-month | 28.33 (4.73)
  3-month: number analyzed (Participants) | 3
  3-month | 31.67 (1.53)

ADVERSE EVENTS:
Time Frame: Client: about 4 months; Caregiver: about 4 months; Volunteer: up to about 16 months (consent through end of funding period)
Description: No adverse events were suspected to be caused by study intervention/procedures.
Groups:
- Experimental: PorchLight Project Intervention Group: Volunteers: Volunteers enrolled undergo the PorchLight project intervention training.
- Experimental: PorchLight Project Intervention Group: Clients: Participants in the intervention group will receive home-based support and respite services from PorchLight Project trained Senior Companion volunteers of the Lutheran Social Services of Minnesota.
- Experimental: PorchLight Project Intervention Group: Caregivers: Caregivers enrolled provide care to a client in the study that receives home-based support and respite services from a PorchLight Project trained Senior Companion volunteer.
Arm/Group | Experimental: PorchLight Project Intervention Group: Volunteers | Experimental: PorchLight Project Intervention Group: Clients | Experimental: PorchLight Project Intervention Group: Caregivers
All-Cause Mortality (participants affected / at risk) | 1/33 | 1/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/7 | 1/4
Other Adverse Events (participants affected / at risk) | 2/33 | 0/7 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: PorchLight Project Intervention Group: Volunteers (N=33) | Experimental: PorchLight Project Intervention Group: Clients (N=7) | Experimental: PorchLight Project Intervention Group: Caregivers (N=4)
Cancer treatment (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fall/ED visit or hospitalization (General disorders) | 0 (0) | 2 (2) | 0 (0)
Transient global amnesia diagnosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: PorchLight Project Intervention Group: Volunteers (N=33) | Experimental: PorchLight Project Intervention Group: Clients (N=7) | Experimental: PorchLight Project Intervention Group: Caregivers (N=4)
Other Adverse Event (General disorders) | 1 | NA | NA — insufficient documentation to categorize further

LIMITATIONS AND CAVEATS:
From PMCID: PMC8127785/PMID: 34036120: "...initial recruitment challenges as well as the COVID-19 pandemic severely curtailed our enrollment of clients and caregivers...Volunteer recruitment was successful (n = 33), and the largest barrier to training completion was early termination related to the pandemic...Due to slower training progress in the rural region, we did not enroll any rural clients or caregivers."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03667924/Prot_SAP_001.pdf
  • Informed Consent Form: Client Assent (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03667924/ICF_002.pdf
  • Informed Consent Form: Caregiver Consent (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03667924/ICF_003.pdf
  • Informed Consent Form: Volunteer Consent (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03667924/ICF_004.pdf
  • Informed Consent Form: Client Consent (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03667924/ICF_005.pdf